CLINICAL TRIAL: NCT03074942
Title: Reslizumab in Patients With Severe Asthma Who Failed to Respond to Omalizumab: a Pilot Study
Brief Title: Reslizumab in Patients With Severe Asthma Who Failed to Respond to Omalizumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEP-RES-2016-01
Record Dates: First submitted 2017-02-28; First posted 2017-03-09 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Severe Asthma
MeSH Terms: conditions — Asthma | interventions — reslizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reslizumab (Experimental): Reslizumab 3 mg/kg once / every 4 weeks during 24 weeks
  Interventions: Drug: Reslizumab

INTERVENTIONS:
Drug: Reslizumab — Reslizumab 3 mg/kg once / every 4 weeks during 24 weeks

SUMMARY:
Approximately, 5% of the patients with asthma suffer a difficult-to-control severe variant of the disease. Despite being treated with inhaled corticosteroids (ICs), long-acting β2-agonists (LABA), oral corticosteroids or omalizumab, one or more components of the control concept (symptoms, exacerbations, bronchial obstruction) remain to be resolved. Omalizumab has been proven to safely reduce asthma exacerbations and to decease symptoms and quality of life in severe allergic asthmatics. However, approximately 25% of the treated patients fail to respond to this monoclonal antibody. The rest of them show different degrees of response, although the rate of asthmatics who achieve control of the disease is unknown because clinical trials of omalizumab have been carried out to assess the impact of the drug on exacerbations, symptoms or even pulmonary function, but its effect on control was not evaluated. Therefore, there is a need to find new therapeutic options for those severe asthmatics who remain uncontrolled despite having received all the recommended therapies (including omalizumab). Reslizumab is a humanized anti-interleukin-5 (IL-5) monoclonal antibody (mAb) that has been recently found to reduce exacerbations and to improve pulmonary function and symptoms in patients with severe asthma and high peripheral eosinophil counts. It would be important to demonstrate that Reslizumab is able to improve the clinical condition of severe asthma patients with no therapeutic options.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 70 years of age,
* Patients diagnosed with severe uncontrolled asthma
* Patients who give informed consent.
* Previous treatment with omalizumab that was discontinued because lack of efficacy (symptoms -ACT <20, exacerbations) or adverse effects.
* Patients with a high blood eosinophil count (400 μl) at least once in the previous 3 years.
* Women should be surgically sterilized, at least 2 years have passed since menopause, or must have a negative pregnancy test within 7 days prior to initiation of treatment.
* Women of childbearing potential (not surgically sterilized or menopausal for less than 2 years) should use a medically accepted method of contraception and should agree to continue using this method during the study and at least 30 days after the end of the study.
* Patient should be willing and able to comply with the study restrictions and attend the visits indicated in the protocol to carry out the follow-up evaluations detailed in the protocol.

Exclusion Criteria:

* Diagnosis of asthma-COPD (Chronic Obstructive Pulmonary Disease) overlap syndrome.
* Active and former smokers of>10 packages / year.
* Exacerbations during the previous 4 weeks.
* Current treatment with omalizumab or last dose of omalizumab in the 5 months prior to inclusion of the patient in the study. 5- Exposure to another monoclonal antibody.
* Participation in another clinical trial.
* Uncontrolled clinically significant disease, which may interfere with study procedures, interpretation of efficacy results, or compromise patient safety.
* Underlying lung disorder.
* Known hypereosinophilic syndrome.
* A pregnant or lactating woman, or who intends to become pregnant during the study.
* Participation in a clinical trial within 30 days prior to the start of treatment.
* Previous exposure to reslizumab or other anti-IL-5 monoclonal antibody.
* Immunodeficiency disorder, including HIV.
* Suspected drug or alcohol abuse.
* Active helminth parasite infection or for which treatment was received in the 6 months prior to the start of treatment.
* History of allergic reaction or hypersensitivity to any component of the study drug.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Asthma Control Test score (ACT) | Baseline and 24 weeks
  Change in Asthma Control Test score (ACT) between baseline and week 24.

SECONDARY OUTCOMES:
Change from baseline in Asthma Control Test (ACT) score | Baseline and 12 weeks
  Change in ACT between baseline and week 12
Change from baseline in the 7-item Asthma Control Questionnaire (ACQ). | Baseline and 24 weeks
  Change in the 7-item ACQ between baseline and week 24.
Percentage of patients that achieve the minimally important difference in ACT | Baseline and 24 weeks
  Percentage of patients that achieve the minimally important difference in ACT (increase of at least 3 ponints) at week 24
Percentage of patients that achieve the minimally important difference in ACQ-7 | Baseline and 24 weeks
  Percentage of patients that achieve the minimally important difference in ACQ-7 (reduction of at least 0.5 ponints) at week 24
Change from baseline in eosinophil count in peripheral blood. | Baseline and 24 weeks
  Change from baseline in eosinophil count in peripheral blood at week 24.
Change from baseline in lung function (FEV1). | Baseline and 24 weeks
  Change from baseline in lung function (FEV1) at week 24.
Number of severe exacerbations of asthma. | 24 weeks
  Number of severe exacerbations of asthma during the 24 weeks of the study.
Change from baseline in the Asthma Quality of Life Questionnaire (AQLQ) score. | Baseline and 24 weeks
  Change from baseline in the AQLQ questionnaire score at week 24.
Change from baseline in exhaled nitric oxide levels. | Baseline and 24 weeks
  Change from baseline in exhaled nitric oxide levels at week 24.
Number of participants with adverse events | 24 weeks
  Number of participants with adverse events
Number of participants with severe adverse events | 24 weeks
  Number of participants with severe adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Luis Pérez de Llano, MD, Study Director — Hospital Universitario Lucus Augusti
Locations (10):
- Spain (10):
  - Hospital Universitari Son Espases, Palma, Balearic Islands
  - Hospital de Sabadell, Sabadell, Barcelona
  - Hospital Universitario de Cruces, Barakaldo, Bizkaia
  - Hospital Galdakao-Usansolo, Galdakao, Vizcaya
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital Reina Sofía, Córdoba
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Universitario La Paz, Madrid
  - Hospital Virgen Del Rocío, Seville
  - Hospital Universitario Dr. Peset, Valencia

IPD SHARING:
Plan to Share IPD: No